CLINICAL TRIAL: NCT03835650
Title: Pelvic Girdle Pain Early Postpartum: Underlying Condition and Associated Factors
Status: Completed | Type: Observational
Sponsor: Żelazna Medical Centre, LLC (Other)
Collaborators: Centre of Postgraduate Medical Education (Other)
Responsible Party: Sponsor
Other Study IDs: PN/19/2019
Record Dates: First submitted 2019-02-04; First posted 2019-02-08 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Pelvic Girdle Pain; Pubic Symphysis Diastasis; Diastasis Recti
MeSH Terms: conditions — Pelvic Girdle Pain; Pubic Symphysis Diastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PGP: Patients in early postpartum period experiencing PGP, confirmed with dedicated functional tests
- no PGP: Patients in early postpartum period, with no symptoms and signs of PGP

SUMMARY:
Background: Pregnancy-related pelvic girdle pain (PGP) can appear during pregnancy, directly after labour or can be delayed to 3 weeks postpartum. Pain is experienced between the posterior iliac crest and the gluteal fold, particularly in the vicinity of the Sacroiliac joints (SIJ). The pain may radiate in the posterior thigh and can also occur in conjunction with/or separately in the symphysis. The endurance capacity for standing, walking, and sitting is diminished. The diagnosis of PGP can be reached after exclusion of lumbar causes. The pain or functional disturbances in relation to PGP must be reproducible by specific clinical tests. Lack of accurate and early diagnosis of the PGP reasons postpartum may contribute to development of chronic condition, lowering quality of life years after delivery.

Objectives: The aim of the project is to evaluate the underlying cause of the severe pelvic girdle pain postpartum (whether it is real PGP or diastasis pubic symphysis) and to assess the differences between females with severe postpartum PGP, mild and moderate PGP and with no PGP in terms of: presence of diastasis pubic symphysis, presence of diastasis recti and linea alba dysfunction, factors associated with labour and maladaptive mental processing (catastrophizing).

Materials and methods: Because of low incidence of researched conditions, a case control study will be the study design of choice. The subjects with PGP will be matched with those with no PGP. Subjects' assessment will consist of palpation and ultrasonography evaluation of diastasis recti(inter-recti distance), ultrasonography assesment of pubic symphysis (inter-pubic width) and mental processing (catastrophizing assessed with Pain Catastrophizing Scale) analysis. Factors connected with labour (time from epidural anaesthesia injection to full dilatation and delivery) will be also investigated.

Expected results: To the investigators' knowledge, postpartum pelvic girdle pain has not been extensively studied so far. The study will bring information about the possible underlying cause of postpartum PGP: whether it is PGP or diastasis pubic symphysis.

ELIGIBILITY:
Inclusion Criteria:

* Natural labour or vacuum extractor or forceps
* for the study group - pain due to PGP confirmed with dedicated functional tests
* for control group with no pain - no pain due to PGP
* agreement to participate

Exclusion Criteria:

* diseases that can mimic PGP f.ex. Scheuermann disease, rheumatoid arthritis, Ehler's-Danlos Syndrome, hip dysplasia
* major peri-partum events like internal haemorrhage, pelvic fracture

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women in early postpartum period (during hospital stay)
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Diastasis Recti: ultrasound measurement of inter-recti distance | one time assessment, during the hospital stay, within 1st week postpartum
  measurement of inter-recti distance (ultrasound assessment at the level of umbilicus, 2cm over the umbilicus and 2 cm below)
Pubic symphysis distance | one time assessment, during the hospital stay, within 1st week postpartum
  assesment of pubic symphysis distance - presence of diastasis pubic symphysis, distance measured by ultrasound

SECONDARY OUTCOMES:
Pain Catastrophizing Scale | one time assessment, during the hospital stay, within 1st week postpartum
  Assesment of Catastrophizing
Epidural anaesthesia | during labour (Time form injection to full cervical dilatation)
  Time form injection to full cervical dilatation
Epidural anaesthaesia2 | during labour (Time form injection to labour)
  Time form injection to labour
Diastasis Recti: inter-recti distance | one time assessment, during the hospital stay, within 1st week postpartum
  measurement of inter-recti distance by palpation examination at the level of umbilicus, 2cm over the umbilicus and 2 cm below

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Postgraduate Medical Education, Warsaw, Masovian Voivodeship, Poland